CLINICAL TRIAL: NCT02262923
Title: Dopamine D-2 Antagonist Use in Poor Responders in IVF: a Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14-0209-A
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2019-03

CONDITIONS: in Vitro Fertilization; Poor Responder
MeSH Terms: interventions — Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Poor responders will be defined as women who have undergone a previous IVF cycle with fewer than 4 oocytes retrieved and at least one of the following two criteria: (1) advanced age (≥40 years) or any other risk factor for poor ovarian response and (2) abnormal ovarian reserve testing (antral follicle count (AFC) < 5-7 or anti-mullerian hormone (AMH) level < 3.6-7.9 pmol/L). Poor responders who will be undergoing a repeat IVF cycle will be recruited for the study with informed consent.
  In the control arm, patients will undergo the same ovarian stimulation protocol as the previous IVF cycle in which they experienced a poor response. Starting 3 weeks prior to the first day of stimulation until the time of ovulation trigger (approximately 5 weeks overall), these patients will receive an oral placebo three times daily.
- Experimental (Experimental): Poor responders will be defined as women who have undergone a previous IVF cycle with fewer than 4 oocytes retrieved and at least one of the following two criteria: (1) advanced age (≥40 years) or any other risk factor for poor ovarian response and (2) abnormal ovarian reserve testing (antral follicle count (AFC) < 5-7 or anti-mullerian hormone (AMH) level < 3.6-7.9 pmol/L). Poor responders who will be undergoing a repeat IVF cycle will be recruited for the study with informed consent.
  In the experimental arm, patients will undergo the same ovarian stimulation protocol as the previous IVF cycle in which they experienced a poor response. Starting 3 weeks prior to the first day of stimulation until the time of ovulation trigger (approximately 5 weeks in total), these patients will receive oral metoclopramide 5mg three times daily..
  Interventions: Drug: metoclopramide

INTERVENTIONS:
Drug: metoclopramide
  Arms: Experimental

SUMMARY:
Metoclopramide is a dopamine D2 receptor antagonist with antiemetic and gastrokinetic properties which has been approved for use in pregnant women. Women with polycystic ovary syndrome (PCOS) have been found to have lower dopaminergic tone and increased ovarian vascularity and vascular endothelial growth factor (VEGF) levels compared to controls. During ovarian stimulation, PCOS patients exhibit greater sensitivity to gonadotropins and increased follicular development. Administration of dopamine D2 antagonists may mimic the low dopaminergic tone noted in PCOS patients, increase VEGF levels, angiogenesis, and subsequently improve follicular growth during ovarian stimulation. This strategy could be used to improve IVF outcomes in poor responders.

The investigators hypothesize that, compared to gonadotropin use alone, the use of metoclopramide in combination with gonadotropins in poor responders undergoing IVF will result in an increased number of mature oocytes obtained at oocyte retrieval and improved IVF outcomes.

DETAILED DESCRIPTION:
Poor responders constitute a significant and challenging population of women to treat with in vitro fertilization (IVF). This population includes women who respond sub-optimally to conventional ovarian stimulation with poor follicular recruitment. The estimated incidence of poor ovarian response ranges from 9-26%. Patients with PCOS are on the opposite end of the spectrum from poor responders. They are often exquisitely sensitive to ovarian stimulation and are predisposed to over-respond with the development of ovarian hyperstimulation syndrome (OHSS). Understanding the underlying mechanisms that enhance their sensitivity may provide insight into the treatment of poor responders. VEGF is a glycoprotein produced by ovarian granulosa cells that enhances vascular permeability and angiogenesis, and has been implicated in the pathogenesis of OHSS. After ovulation is triggered by LH or hCG, follicular expression of VEGF increases, which is crucial for corpus luteum function and steroidogenesis. However, excessive VEGF production can lead to third-space shifts of fluids, ascites, and other life-threatening features of OHSS. Serum concentrations and granulosa cell expression of VEGF have been shown to be higher in women with PCOS than in controls. Interestingly, compared with controls, patients with PCOS have also been shown to have lower levels of the neurotransmitter dopamine and dopamine D2 receptor levels in the ovary. Administration of dopamine D2 agonists has been shown in animal and human studies to decrease ovarian VEGF production and reduce the risk of OHSS. In this study, the investigators propose a novel approach of administering a dopamine D2 antagonist to poor responders to mimic the low dopaminergic tone of PCOS patients, with the goal of increasing VEGF production and follicular development during ovarian stimulation. Metoclopramide is a dopamine D2 antagonist with antiemetic and prokinetic properties and an established safety profile in pregnancy. The investigators hypothesis is that metoclopramide use prior to, and in conjunction with, conventional gonadotropin stimulation can improve IVF outcomes in poor responders.

ELIGIBILITY:
Inclusion Criteria:

* Poor responders undergoing a repeat IVF cycle defined as women who have undergone at least one previous IVF cycle with fewer than 4 oocytes retrieved and at least one of the following:

  * Advanced age (≥40 years) or any other risk factor for poor ovarian response
  * Abnormal ovarian reserve testing (antral follicle count (AFC) < 5-7 or anti-mullerian hormone (AMH) level < 3.6-7.9 pmol/L)

Exclusion Criteria:

* Subjects who have previously been recruited into this study and either had cycle cancellation, underwent retrieval or dropped out of the study.
* Women with contraindications or allergies to metoclopramide.
* Women with elevated prolactin levels or known to have pituitary microadenomas or macroadenoma.
* Women who are taking dopamine agonist medications.

Ages: 21 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 1 year

SECONDARY OUTCOMES:
Number of mature follicles (≥1.5cm) seen on transvaginal ultrasound at the time of ovulation trigger | 1 year
Peak serum estradiol levels measured at the time of ovulation trigger shot | 1 year
Ratio of mature/ immature oocytes obtained at oocyte retrieval | 1 year
Follicular fluid levels of VEGF, VEGFR-1 and VEGFR-2 | 1 year
Total dose of gonadotropins used and number of days of stimulation | 1 year
Fertilization rates | 1 year
Number of embryos on day 3 and 5 | 1 year
Pregnancy and implantation rates | 1-2 years
Serum prolactin levels on cycle day 3,7 and at the time of ovulation trigger | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada